CLINICAL TRIAL: NCT03762278
Title: Can Supplemental Leucine Offset Disuse-induced Muscle Atrophy?
Acronym: LEU-DIMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: RG_16-206
Record Dates: First submitted 2017-02-20; First posted 2018-12-03 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2018-11

CONDITIONS: Muscle Disuse Atrophy
Keywords: Unilateral Immobilisation; Leucine; Muscle Wasting; Nutritional Intervention
MeSH Terms: conditions — Muscular Disorders, Atrophic; Muscular Atrophy | interventions — Leucine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Immobilised leg and leucine (Experimental): Participants consuming leucine supplementation with measures obtained from the uni-laterally immobilised leg.
  Interventions: Dietary Supplement: Leucine
- Non-immobilised leg and leucine (Active Comparator): Participants consuming leucine supplementation with measures obtained from the non-immobilised leg.
  Interventions: Dietary Supplement: Leucine
- Immobilised leg and placebo (Placebo Comparator): Participants consuming placebo supplementation with measures obtained from the uni-laterally immobilised leg.
  Interventions: Dietary Supplement: Placebo
- Non-immobilised leg and placebo (Placebo Comparator): Participants consuming placebo supplementation with measures obtained from the non-immobilised leg.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Leucine — Participants will ingest 15g of leucine supplementation/day during the immobilisation period. Leucine supplementation will be administered in powdered form (Infinit Nutrition, Canada) and participants will be required to consume 5g of leucine mixed with 250-300 ml of water during each meal. Leucine is a dietary supplement according to the US FDA. This supplementation protocol has been demonstrated in humans (Murphy et al., 2016, AJCN) with no reported side effects. The quantity of leucine supplementation falls well within the safe limits outlined by Rasmussen et al. (2016). Infinit Nutrition Leucine is in compliance with banned substances requirements as espoused by the World Anti-Doping Agency. Infinit Nutrition Leucine is not a medicinal product.
  Other Names: Infinit Nutrition Leucine
  Arms: Immobilised leg and leucine; Non-immobilised leg and leucine
Dietary Supplement: Placebo — Participants will ingest 15g of placebo supplementation/day during the immobilisation period. Placebo supplementation will be administered in powdered form and participants will be required to consume 5g of placebo supplementation mixed with 250-300 ml of water during each meal (3x/day).
  Placebo supplementation will contain 5g of non-essential amino acids (Infinit Nutrition, Canada) and will be calorically matched to the leucine supplementation.This supplementation protocol has been demonstrated previously in humans, with no reported side effects (Murphy et al., 2016, AJCN).
  Other Names: Infinit Nutrition Placebo
  Arms: Immobilised leg and placebo; Non-immobilised leg and placebo

SUMMARY:
Ageing is associated with a gradual decline in muscle mass that is detrimental to both physical function and metabolic health, increasing the risk of morbidity and mortality. The loss of protein muscle mass with ageing is poorly understood, but it may partly relate to inactivity/disuse (i.e. during injury or hospitalization). Periods of inactivity/disuse blunt the ability of muscle to grow (termed anabolic blunting), leading to a loss of muscle mass and strength. An accumulation of these periods over a lifetime promotes the devastating loss of muscle protein mass and strength seen with ageing.

Disuse-induced muscle loss is underpinned by a blunted muscle anabolic response to protein nutrition. Supplementing the diet with the amino acid leucine may offer a potential solution to alleviate muscle mass and strength loss during disuse. In fact, leucine is suggested to promote muscle protein growth and reduce muscle protein loss during disuse in rats, but this is yet to be shown in humans. Accordingly, the proposed study will investigate whether leucine supplementation can offset muscle and strength loss during short-term disuse.

Twenty-four healthy (non-obese, non-diabetic, non-smokers) men aged 18-35 years will initially complete a lower-limb strength assessment and undergo a body composition scan three days later. The following morning, participants will be randomly assigned to ingest either 5g of leucine (n=12) or a caloric-matched placebo (n=12) with each meal over a 7 d period of a single-leg immobilisation. Immediately following immobilisation participants will undergo another body composition scan. Additionally, a stable isotope infusion will be combined with serial muscle biopsies from the thigh of each leg to determine the measure rates of muscle protein synthesis in the fasted state and in the 'early' and 'late' phase of feeding. A day later, the assessment of muscle strength will be repeated.

DETAILED DESCRIPTION:
It is well established that skeletal muscle mass progressively declines with healthy ageing, a phenomenon commonly termed sarcopenia. Overtime, this leads to a loss in functional independence and provides an increased risk of developing a co-morbidity. Recent estimates suggest that 30% of those aged 75-84 years suffer from sarcopenia. As the 85-and-over population are rapidly expanding, sarcopenia places a considerable socio-economic burden to healthcare services. From a physiological perspective, the maintenance of muscle mass is dependent on a fine balance between muscle protein synthesis (MPS) and breakdown (MPB) rates. In old age, the MPS response to nutrition is impaired (termed 'anabolic resistance'), leaving muscle in a chronic catabolic state and ultimately underpinning the progression of sarcopenia.

Age-associated muscle anabolic resistance may stem from an accumulation of periods of inactivity/disuse, which are strongly associated with a decline in muscle mass (atrophy) in both the young and old. In fact, the associated loss of muscle mass is the most rapid at the onset of muscle disuse, with significant declines in muscle mass occurring after just 5 days of disuse. This is of particular importance since the average length of hospitalization in older individuals in 5-6 days. Disuse-induced muscle deconditioning is attributed to declines in MPS in response to nutrition, and potentially an elevated MPB. Therefore, an accumulation of these periods of disuse over a lifetime may lead to an acceleration in the trajectory of sarcopenia that is commonly seen with ageing. Consequently, nutritional strategies to maximize healthy musculoskeletal ageing should focus on alleviating muscle metabolic dysregulation during short-term disuse.

One approach to counteract muscle deterioration during short-term disuse is to increase dietary protein consumption. In fact, adequate protein intake is a necessity for muscle to remain in a positive net protein balance, with the importance of this nutritional intervention increasing during periods of disuse. However, this approach is not always feasible as activity levels are more limited during periods of disuse and individuals are thus less likely to consume adequate nutritional intake. A more feasible approach may be to enhance the anabolic potency of sub-optimal protein doses through supplementation with the amino acid, leucine. Leucine is unique in its ability to increase the protein balance more so than any other amino acid through stimulation of MPS and suppression of MPB. Leucine provides a strong anti-catabolic effect during hind limb immobilization in rats, which has yet to be examined in humans. Therefore, it is clear that leucine represents a viable strategy to offset the dysregulation of MPS and MPB and preserve musculoskeletal health during short-term disuse in both young and old individuals and thus warrants further investigation.

Participants:

Twenty-four healthy (non-obese, non-diabetic, non-smokers) males aged 18-35 years will be recruited to participate in the study. The current study will be a placebo controlled double-blind study with two intervention groups, in which, participants will be randomly assigned to receive supplemental leucine (LEU; n=12) or placebo (PLA; n=12) during 7 days of unilateral leg immobilization. Participants will be active, but athletically untrained (i.e. exercise ≤3x/week). All study procedures will be clearly explained and participants will provide written informed consent prior to obtaining baseline measures.

Enrolment:

Participants will be invited to the University of Birmingham's School of Sport, Exercise and Rehabilitation Sciences. Upon arrival, a researcher involved in the trial will explain the study design and interventions to the participant. Participants will be given the opportunity to ask any questions related to the study and will be given time to decide whether or not to take part. If the participant is happy to take part the participant will be asked to sign a consent form and fill in a health questionnaire. When the participant has left, the participant will be categorized at random to the leucine or placebo group. Participants will be asked to fill in a three-day diet diary to assess habitual dietary intake.

Preliminary assessments:

Following explanation of the study and the acquisition of informed consent, participants will report to the laboratory at 0800-0900h having fasted for 10 hours and refrained from vigorous exercise and alcohol for 24 hours previously. Participants baseline muscle function will be acquired through measures of maximal isometric and isokinetic strength of the knee extensor and flexor muscles using an isokinetic dynamometer. Following strength testing the investigators will provide individuals with a three-day diet diary and activity monitor. Three days following the baseline strength measures, participants will once again report to the laboratory at 0800-0900h following a 10h overnight fast. Participants will be weighed on a digital scale to the nearest 0.1kg in light clothing. Dual x-ray absorptiometry (DXA) and ultrasound scans will be conducted to determine the composition of the thigh (fat and fat free mass).

Immobilization:

At 0800-0900h on the morning following preliminary assessments, participants will undergo 7 days of unilateral leg immobilization. A single leg will be randomly selected (counterbalanced left/right) and placed in a full-leg knee brace. Participants will ambulate using crutches and perform daily ankle exercises to minimize the risk of deep vein thrombosis, as indicated by a qualified physiotherapist. Participants will also be permitted to remove the knee brace during overnight sleep. A trained physiotherapist will instruct the participant on the safe use of crutches (i.e climbing stairs). During each main meal in the immobilization period, participants will consume 5 g of a powdered LEU or PLA supplement with 250-300 ml of water, which is within the safe limits. Dietary intake will be controlled throughout the immobilization period according to the individuals total calorie intake (derived from standardized equations), with a macro-nutrient composition of 55% carbohydrate, 30% fat and 15% protein. The total quantity of protein ingestion will equate to 1.0g/kg/day. Participant's activity levels will be monitored throughout the 7 day period through a wrist-worn activity monitor.

Experimental trials:

On the morning marking the end of the 7 d immobilization period participants will report to the laboratory at 0600-0700h following an overnight fast. Ultrasound and DXA assessments will be repeated, immediately after which a catheter will be inserted into a forearm vein of both arms for i) frequent blood sampling at -150, -90, 0, 20, 40, 60, 80, 120, 180, 240-minutes of the experimental trial (∼100mL in total) and ii) a continuous infusion of a stable isotope amino acid tracer (L- [ring] 13C6 phenylalanine). Participants will remain in a supine position throughout the trial. After 150 min of infusion, a muscle biopsy will be obtained from the quadriceps muscle of immobilized and non-immobilized legs under local anaesthetic. Participants will then consume a 20g milk protein beverage. Further biopsies will be obtained from both legs after 270-min and 390-mins of infusion. Thus, a total of 6 invasive muscle biopsies will be obtained during the trial (3 from each leg), with each biopsy obtained from a separate incision spaced ∼3cm apart. This two- stage stable-isotope infusion design allows efficient assessment of MPS in the transition from post-absorptive (0-120 min) to postprandial conditions (120-240 min). Leg strength will be reassessed a day following the stable isotope infusion at 0800-0900h following a 10 hr fast to avoid any interference effect of prior contraction on muscle protein turnover.

Data Analysis:

To calculate myofibrillar and mitochondrial protein synthesis, the investigators will adopt typical sophisticated mass spectrometry techniques to determine isotopic tracer enrichment in biopsy-isolated muscle proteins and plasma. Intramuscular "anabolic signals" (in the mTORC1 pathway) and "catabolic" signals will be determined via western blot and q-rtPCR analysis. High resolution respirometry will also be used to assess the mitochondrial function of biopsy-isolated skeletal muscle tissue in both the control and immobilized limbs.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-35 years old
2. Sex: male
3. BMI: 18-25 kg/m2
4. Diagnosis and general health: Good general health defined as (i) no known cardiovascular or metabolic disease, ii) non-smokers, iii) accustomed to normal levels of physical activity
5. Compliance: understands and is willing, able and likely to comply with all study procedures and restrictions.
6. Consent: demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent

Exclusion Criteria:

1. Health problems such as: i) heart disease, ii) rheumatoid arthritis, iii) diabetes, iv) poor lung function, v) uncontrolled hypertension, vi) lactose intolerance or viI) any health conditions that might put the participant at risk for this study.
2. Family history of thrombosis
3. Involvement in regular structured exercise (resistance or endurance) training at the time of the study.
4. Regular consumption of any analgesic or anti-inflammatory drug(s), either prescription or non-prescription
5. Taking any medications known to affect protein metabolism (e.g. b-blockers, corticosteroids, non-steroidal anti- inflammatories, or prescription strength acne medications). Additional medications and/or supplementation aids (e.g. whey protein) will be deemed inappropriate based on the PI's discretion.
6. Daily protein intake; individuals with protein intake that equates to <0.8 or >1.2 g/kg/day will be excluded from the proposed study, as altering the daily protein intake of individuals drastically over the 7 day period is expected to significantly impact muscle protein metabolism independent of the supplementation and/or immobilisation protocol.
7. Infused with a stable isotope within 3 years prior to study participation

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants must be male.
Enrollment: 24 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
The change in the lean mass of the leg muscles following the 7 day immobilisation period. | At baseline and then 7-days following the onset of immobilisation
  The change in the lean mass of the leg muscles following the 7 day immobilisation period.

SECONDARY OUTCOMES:
The rates of post-absorptive and post-prandial myofibrillar protein synthesis response to 20 g of milk protein after a 7 day period of disuse. | After 7 days of single-leg immobilisation in both the immobilised and non-immobilised leg
  The rates of post-absorptive and post-prandial myofibrillar protein synthesis response to 20 g of milk protein after a 7 day period of disuse.

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Breen, PhD, Principal Investigator — University of Birmingham
Locations (1):
- University of Birmingham, School of Sport, Exercise and Rehabilitation Sciences, Edgbaston, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Edwards SJ, Smeuninx B, Mckendry J, Nishimura Y, Luo D, Marshall RN, Perkins M, Ramsay J, Joanisse S, Philp A, Breen L. High-dose leucine supplementation does not prevent muscle atrophy or strength loss over 7 days of immobilization in healthy young males. Am J Clin Nutr. 2020 Nov 11;112(5):1368-1381. doi: 10.1093/ajcn/nqaa229. PMID 32910813